CLINICAL TRIAL: NCT06553651
Title: Necrosectomy With Cryotechnology for Accelerated Removal
Acronym: NECTAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher C. Thompson, MD, MSc (Other)
Collaborators: Erbe Elektromedizin GmbH (Industry)
Responsible Party: Sponsor-Investigator, Christopher C. Thompson, MD, MSc, Director of Endoscopy, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P002218
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Necrosis; Acute Pancreatitis; Acute Pancreatic Necrosis; Necrosis; Necrosis Pancreas; Walled-Off Pancreatic Necrosis
Keywords: Direct Endoscopic Necrosectomy (DEN); Endoscopic Necrosectomy; Pancreatic Necrosectomy; Necrosectomy; Cryotherapy; Cryotechnology
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Pancreatitis; Necrosis | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Pilot, single-center, open-label, prospective, single-arm clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cryotechnology Necrosectomy Procedure (Experimental): Enrolled subjects will undergo direct endoscopic necrosectomy using 1.7 mm single use, flexible cryoprobes, aimed at effectively removing necrotic tissue within the pancreatic cavity.
  Interventions: Device: Cryotechnology Necrosectomy Procedure

INTERVENTIONS:
Device: Cryotechnology Necrosectomy Procedure — Subjects undergo necrosectomy with 1.7 mm flexible cryoprobes, either concurrently with stent placement or post-placement, at the Investigator's discretion. The cryoprobe will freeze the necrotic tissue and extracted en-bloc. A maximum of 4 cryotechnology procedures will be performed, with each procedure aiming for significant debris removal and clinical improvement of walled-off pancreatic necrosis (WOPN) symptoms.
  Other Names: Cryotherapy

SUMMARY:
Pancreatic necrosis is a serious complication of acute pancreatitis. Pancreatic necrosis involves the irreversible death of pancreatic tissue, which can lead to severe health issues, including infections and an increased risk of death. An endoscopic procedure called direct endoscopic necrosectomy (DEN) is typically performed to remove this necrotic pancreatic tissue as a minimally invasive treatment. This procedure is performed using a thin, flexible, lighted tube called an endoscope and endoscopic instruments that are used with working channels through the scope. Current methods for removing necrotic tissue involve using endoscopic devices such as snares, baskets, nets, and forceps. However, these standard methods are often not very effective because the necrotic tissue can be sticky and hard to grasp. This DEN procedure is part of regular clinical care to treat this condition and remove necrotic tissue from the pancreas.

For this research study, the same DEN procedure will be followed with the exception of the device used for the removal of the necrotic tissue. Instead of using forceps, snares, or other traditional tools, a cryoprobe will be used. Cryoprobes work by using extremely cold temperatures to freeze and adhere to the necrotic tissue, making it easier to remove. This method might be better because it can secure larger tissue samples and potentially reduce complications associated with traditional methods. Cryotechnology is successfully used in endoscopy to remove necrotic tissue, foreign bodies and more, but has not been extensively tested in pancreatic necrosis. Cryoprobes are FDA approved medical devices with an established safety record. They are used successfully in very sensitive areas such as the lungs. This study aims to evaluate the safety and effectiveness of cryotechnology for DEN.

DETAILED DESCRIPTION:
Acute pancreatitis is the most common gastrointestinal disease requiring acute hospital admission. Pancreatic necrosis, a serious complication of acute pancreatitis, is the irreversible death of pancreatic tissue and, in some cases, surrounding abdominal tissue. Worldwide, the incidence of acute pancreatitis ranges from 13 to 45 cases per 100,000 people per year, with a subset progressing to necrotizing pancreatitis. Approximately 5-10% of acute pancreatitis cases progress to this severe form, which carries a significant morbidity and mortality burden, with mortality rates escalating to as high as 32% in cases complicated by infection. The management of pancreatic necrosis is challenging and requires several therapeutic interventions to mitigate the high morbidity and mortality associated with this condition.

The treatment of pancreatic necrosis includes several therapeutic strategies, each with varying degrees of invasiveness, efficacy, and associated risks:

Surgical debridement: Traditionally, surgical debridement has been the cornerstone of treatment for pancreatic necrosis, with the goal of removing necrotic tissue. Although effective, this approach is associated with significant risks, including high morbidity and mortality rates, as high as 39% in some studies. Surgical debridement is a very invasive procedure and often not suitable for patients with severe pancreatitis and their often compromised health status.

Percutaneous Catheter Drainage (PCD): A less invasive alternative to surgery, PCD facilitates drainage of infected necrotic fluid collections. However, its effectiveness is limited by its inability to effectively remove solid necrotic debris. This limitation often requires additional interventions or procedures.

Endoscopic necrosectomy: This minimally invasive technique involves the endoscopic removal of necrotic tissue through the stomach or duodenum. Endoscopic necrosectomy, particularly when used in a step-up approach that may combine PCD with endoscopic drainage and debridement, has been shown to reduce morbidity compared to surgery. Despite the better outcome of the endoscopic technique, there is a gap in effective devices for necrotic tissue removal. Primarily, devices that are utilized include polypectomy snares, biliary baskets, food bolus nets (Roth nets), and forceps. As they are not designed for this indication, their use is often sophisticated and not always successful. As a result, fragmentation and removal as well as a complete debridement of the necrotic tissue is not always achieved, and multiple sessions are required. In a large multicenter trial in the United States, the total number of interventions ranged from 3.1 (immediate direct endoscopic necrosectomy DEN) to 3.9 (delayed DEN). This reflects a significant limitation in the current management of pancreatic necrosis and requires alternative approaches.

Cryotechnology:

In contrast to conventional methods, cryotechnology provides a method for obtaining large tissue samples by utilizing the Joule-Thompson effect for the production of extremely cold temperatures at the probe tip.This involves the internal flow of carbon dioxide (CO2) from a high pressure source to a small nozzle at the tip of the instrument where it expands. The gas expansion causes a large temperature drop (Joule-Thomson effect) and as a result, the surrounding instrument tip is cooled. The expanded gas is returned internally from the tip to the cryosurgical unit via the return tube.

This technology is widely available and used in endoscopy, particularly in the field of pulmonology. Cryoprobes are flexible endoscopic instruments that are currently available in different diameters, 1.1 mm, 1.7 mm, and 2.4 mm. The longstanding safety and efficacy profile have demonstrated results in the safe and efficient management of the following clinical applications, biopsy, extraction and devitalization. They are intended for applications such as the removal of foreign bodies, mucus plugs, blood clots, necrotic tissue, tissue tumors (palliative recanalization) and tissue biopsies. Tissue samples obtained with this technique (cryoadhesion) have been shown to be heavier and larger than those obtained with conventional forceps.

Potential for Pancreatic Necrosis and Significance:

The successful implementation of cryotechnology for extraction suggests its potential applicability for pancreatic necrosectomy. The use of cryoprobes for minimally invasive endoscopic removal of necrotic pancreatic tissue may represent a novel approach that overcomes the limitations of existing strategies. The ability of cryotechnology to secure larger tissue samples without significant bleeding risks, coupled with its safety profile, provides an opportunity to improve the management of necrotizing pancreatitis. This study aims to investigate the safety, efficacy, and feasibility of cryoprobe use for the endoscopic removal of necrotic tissue, setting the stage for future clinical advances in the management of necrotizing pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years and above, inclusive of both males and females.
* Patients with symptomatic pancreatic necrosis resulting from acute pancreatitis, indicated for endoscopic necrosectomy following endoscopic ultrasound (EUS)-guided drainage.
* Imaging indicative of ≥30% necrotic material within the pancreas.
* Walled-off pancreatic necrosis (WOPN) size ≥6 cm.
* Subjects able to tolerate repeated endoscopic procedures.
* Capacity for providing informed consent.
* Understanding of study requirements, provision of written informed consent, and willingness and ability to attend required follow-up assessments through 21 (+/- 7) days.

Exclusion Criteria:

* Inability to provide informed consent.
* Unwillingness to undergo repeated endoscopies.
* Presence of documented Pseudoaneurysm > 1cm within the WOPN.
* Intervening gastric varices or unavoidable blood vessels within the access tract.
* Use of dual antiplatelet therapy or therapeutic anticoagulation that cannot be temporarily discontinued.
* Any condition deemed by the investigator to compromise the safety of undergoing an endoscopic procedure.
* Pregnancy, lactation, or absence of reliable contraception in women of childbearing potential.
* Current enrollment in another investigational trial with potential to interfere with this study's endpoint analyses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Technical Success Rate | Baseline, Follow-up Visit Day 21
  To evaluate the effectiveness of cryotechnology for the removal of necrotic pancreatic tissue. Achievement of at least 70% removal of necrotic debris from the pancreatic collection being treated, as determined by change in computed tomography (CT) evaluation from baseline to 21 days post-treatment.

SECONDARY OUTCOMES:
Safety and Procedure-Related Adverse Events | Procedure Day 0, Follow-up Visit Day 21
  To assess the safety profile of using cryotechnology for necrosectomy by monitoring the incidence of intraprocedure-related adverse events, including intracaviteal bleeding during the procedure, aspiration, septic event, and perforation, through follow-up day 21.
Mean Total Procedure Time | Procedure Day 0, Reintervention (if needed)
  To determine the efficiency of cryotechnology for necrosectomy by measuring the mean total procedure time required to achieve at least a 70% reduction in necrosis. Time from first insertion of the cryoprobe into the endoscope to the end of its use (last extraction from the endoscope). The total procedure time for achieving clearance of necrosis will be assessed across all necrosectomy sessions for each patient.
Total Number of Reinterventions | From Procedure Day 0 through Follow-up Visit Day 21
  To quantify the necessity for additional interventions by recording the total number of reinterventions per patient required to achieve treatment success.
Clinical Improvement within 72 Hours | Baseline, Procedure Day 0, up to 3 days post-procedure
  To evaluate early clinical improvement, defined as observable patient recovery within 72 hours following the index intervention, improvement in Gastrointestinal Symptom Rating Scale (GSRS) and improvement in c-reactive protein (CRP) labs from baseline. GSRS is seven-point Likert-type scale with 1 being no symptoms, to 7 being worst possible symptoms.
Duration of Hospital Stay | From Procedure Day 0 through date of discharge
  To assess the impact of cryotechnology on the length of hospital stay, measured from the index intervention to discharge in days.
Quality of Life (QOL) | Baseline, Follow-up Day 21
  Evaluate QoL improvement using the 12 question Short Form survey (SF-12) scores from baseline to 21 (+/- 7) days post-last cryo debridement. Scores range from 0-100. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C. Thompson, MD, MSc, Principal Investigator — Brigham and Womens Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will be shared on a case by case basis with an Institutional data transfer agreement in place.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 12 months after publication
Access Criteria: IPD requests should be made directly to the PI who will determine feasibility of the request. Institutional data transfer agreement will need to be executed to share data.

REFERENCES:
- [Background] Arvanitakis M, Dumonceau JM, Albert J, Badaoui A, Bali MA, Barthet M, Besselink M, Deviere J, Oliveira Ferreira A, Gyokeres T, Hritz I, Hucl T, Milashka M, Papanikolaou IS, Poley JW, Seewald S, Vanbiervliet G, van Lienden K, van Santvoort H, Voermans R, Delhaye M, van Hooft J. Endoscopic management of acute necrotizing pancreatitis: European Society of Gastrointestinal Endoscopy (ESGE) evidence-based multidisciplinary guidelines. Endoscopy. 2018 May;50(5):524-546. doi: 10.1055/a-0588-5365. Epub 2018 Apr 9. PMID 29631305
- [Background] Yadav D, Lowenfels AB. The epidemiology of pancreatitis and pancreatic cancer. Gastroenterology. 2013 Jun;144(6):1252-61. doi: 10.1053/j.gastro.2013.01.068. PMID 23622135
- [Background] Trikudanathan G, Wolbrink DRJ, van Santvoort HC, Mallery S, Freeman M, Besselink MG. Current Concepts in Severe Acute and Necrotizing Pancreatitis: An Evidence-Based Approach. Gastroenterology. 2019 May;156(7):1994-2007.e3. doi: 10.1053/j.gastro.2019.01.269. Epub 2019 Feb 15. PMID 30776347
- [Background] Pinto S, Bellizzi S, Badas R, Canfora ML, Loddo E, Spada S, Khalaf K, Fugazza A, Bergamini S. Direct Endoscopic Necrosectomy: Timing and Technique. Medicina (Kaunas). 2021 Nov 28;57(12):1305. doi: 10.3390/medicina57121305. PMID 34946249
- [Background] Bang JY, Lakhtakia S, Thakkar S, Buxbaum JL, Waxman I, Sutton B, Memon SF, Singh S, Basha J, Singh A, Navaneethan U, Hawes RH, Wilcox CM, Varadarajulu S; United States Pancreatic Disease Study Group. Upfront endoscopic necrosectomy or step-up endoscopic approach for infected necrotising pancreatitis (DESTIN): a single-blinded, multicentre, randomised trial. Lancet Gastroenterol Hepatol. 2024 Jan;9(1):22-33. doi: 10.1016/S2468-1253(23)00331-X. Epub 2023 Nov 18. PMID 37980922
- [Background] van Brunschot S, Hollemans RA, Bakker OJ, Besselink MG, Baron TH, Beger HG, Boermeester MA, Bollen TL, Bruno MJ, Carter R, French JJ, Coelho D, Dahl B, Dijkgraaf MG, Doctor N, Fagenholz PJ, Farkas G, Castillo CFD, Fockens P, Freeman ML, Gardner TB, Goor HV, Gooszen HG, Hannink G, Lochan R, McKay CJ, Neoptolemos JP, Olah A, Parks RW, Peev MP, Raraty M, Rau B, Rosch T, Rovers M, Seifert H, Siriwardena AK, Horvath KD, van Santvoort HC. Minimally invasive and endoscopic versus open necrosectomy for necrotising pancreatitis: a pooled analysis of individual data for 1980 patients. Gut. 2018 Apr;67(4):697-706. doi: 10.1136/gutjnl-2016-313341. Epub 2017 Aug 3. PMID 28774886
- [Background] Mohamadnejad M, Anushiravani A, Kasaeian A, Sorouri M, Djalalinia S, Kazemzadeh Houjaghan A, Gaidhane M, Kahaleh M. Endoscopic or surgical treatment for necrotizing pancreatitis: Comprehensive systematic review and meta-analysis. Endosc Int Open. 2022 Apr 14;10(4):E420-E428. doi: 10.1055/a-1783-9229. eCollection 2022 Apr. PMID 35433210
- [Background] American Society for Gastrointestinal Endoscopy Technology Committee; Saumoy M, Trindade AJ, Bhatt A, Bucobo JC, Chandrasekhara V, Copland AP, Han S, Kahn A, Krishnan K, Kumta NA, Law R, Obando JV, Parsi MA, Trikudanathan G, Yang J, Lichtenstein DR; American Society for Gastrointestinal Endoscopy Technology Committee Chair. Summary: endoscopic therapies for walled-off necrosis. Gastrointest Endosc. 2023 Jun;97(6):1001-1002. doi: 10.1016/j.gie.2023.02.008. Epub 2023 Apr 26. No abstract available. PMID 37115165
- [Background] van Santvoort HC, Besselink MG, Bakker OJ, Hofker HS, Boermeester MA, Dejong CH, van Goor H, Schaapherder AF, van Eijck CH, Bollen TL, van Ramshorst B, Nieuwenhuijs VB, Timmer R, Lameris JS, Kruyt PM, Manusama ER, van der Harst E, van der Schelling GP, Karsten T, Hesselink EJ, van Laarhoven CJ, Rosman C, Bosscha K, de Wit RJ, Houdijk AP, van Leeuwen MS, Buskens E, Gooszen HG; Dutch Pancreatitis Study Group. A step-up approach or open necrosectomy for necrotizing pancreatitis. N Engl J Med. 2010 Apr 22;362(16):1491-502. doi: 10.1056/NEJMoa0908821. PMID 20410514
- [Background] Besselink MG, van Santvoort HC, Nieuwenhuijs VB, Boermeester MA, Bollen TL, Buskens E, Dejong CH, van Eijck CH, van Goor H, Hofker SS, Lameris JS, van Leeuwen MS, Ploeg RJ, van Ramshorst B, Schaapherder AF, Cuesta MA, Consten EC, Gouma DJ, van der Harst E, Hesselink EJ, Houdijk LP, Karsten TM, van Laarhoven CJ, Pierie JP, Rosman C, Bilgen EJ, Timmer R, van der Tweel I, de Wit RJ, Witteman BJ, Gooszen HG; Dutch Acute Pancreatitis Study Group. Minimally invasive 'step-up approach' versus maximal necrosectomy in patients with acute necrotising pancreatitis (PANTER trial): design and rationale of a randomised controlled multicenter trial [ISRCTN13975868]. BMC Surg. 2006 Apr 11;6:6. doi: 10.1186/1471-2482-6-6. PMID 16606471
- [Background] Yachimski P, Landewee CA, Campisano F, Valdastri P, Obstein KL. The waterjet necrosectomy device for endoscopic management of pancreatic necrosis: design, development, and preclinical testing (with videos). Gastrointest Endosc. 2020 Sep;92(3):770-775. doi: 10.1016/j.gie.2020.04.024. Epub 2020 Apr 22. PMID 32334018
- [Background] Yan L, Dargan A, Nieto J, Shariaha RZ, Binmoeller KF, Adler DG, DeSimone M, Berzin T, Swahney M, Draganov PV, Yang DJ, Diehl DL, Wang L, Ghulab A, Butt N, Siddiqui AA. Direct endoscopic necrosectomy at the time of transmural stent placement results in earlier resolution of complex walled-off pancreatic necrosis: Results from a large multicenter United States trial. Endosc Ultrasound. 2019 May-Jun;8(3):172-179. doi: 10.4103/eus.eus_108_17. PMID 29882517
- [Background] Giri M, Huang G, Puri A, Zhuang R, Li Y, Guo S. Efficacy and Safety of Cryobiopsy vs. Forceps Biopsy for Interstitial Lung Diseases, Lung Tumors, and Peripheral Pulmonary Lesions: An Updated Systematic Review and Meta-Analysis. Front Med (Lausanne). 2022 Mar 10;9:840702. doi: 10.3389/fmed.2022.840702. eCollection 2022. PMID 35372452
- [Background] Wirsing L, Linzenbold W, Jaeger SU, Stahl P, Ott G, Leibold T, Enderle M, Albert J, Peveling-Oberhag J. A new tool for bile duct tissue sampling: ex vivo clinical evaluation of intraductal cryobiopsy for cholangioscopy. Endosc Int Open. 2022 Jun 10;10(6):E809-E814. doi: 10.1055/a-1797-8966. eCollection 2022 Jun. PMID 35692925
- [Background] Klein JT, Berger F, Linzenbold W, Jager L, Enderle MD, Bosmuller H, Mundhenk J, Schwentner C, Bolenz C. Cryobiopsy in the Upper Urinary Tract: Preclinical Evaluation of a Novel Device. Urology. 2019 Jan;123:273-279. doi: 10.1016/j.urology.2018.10.003. Epub 2018 Oct 9. PMID 30312669
- [Background] Behr J, Gunther A, Bonella F, Dinkel J, Fink L, Geiser T, Geissler K, Glaser S, Handzhiev S, Jonigk D, Koschel D, Kreuter M, Leuschner G, Markart P, Prasse A, Schonfeld N, Schupp JC, Sitter H, Muller-Quernheim J, Costabel U. S2K Guideline for Diagnosis of Idiopathic Pulmonary Fibrosis. Respiration. 2021;100(3):238-271. doi: 10.1159/000512315. Epub 2021 Jan 22. PMID 33486500
- [Background] Aboudara M, Maldonado F. Transbronchial cryobiopsy for diffuse parenchymal lung diseases: evidence that demands a (favorable) verdict. Ann Transl Med. 2020 Oct;8(20):1324. doi: 10.21037/atm-20-2995. No abstract available. PMID 33209904
- [Background] Hetzel J, Eberhardt R, Herth FJ, Petermann C, Reichle G, Freitag L, Dobbertin I, Franke KJ, Stanzel F, Beyer T, Moller P, Fritz P, Ott G, Schnabel PA, Kastendieck H, Lang W, Morresi-Hauf AT, Szyrach MN, Muche R, Shah PL, Babiak A, Hetzel M. Cryobiopsy increases the diagnostic yield of endobronchial biopsy: a multicentre trial. Eur Respir J. 2012 Mar;39(3):685-90. doi: 10.1183/09031936.00033011. Epub 2011 Aug 18. PMID 21852332
- [Background] Herth FJ, Mayer M, Thiboutot J, Kapp CM, Sun J, Zhang X, Herth J, Kontogianni K, Yarmus L. Safety and Performance of Transbronchial Cryobiopsy for Parenchymal Lung Lesions. Chest. 2021 Oct;160(4):1512-1519. doi: 10.1016/j.chest.2021.04.063. Epub 2021 May 7. PMID 33971147
- [Background] Peveling-Oberhag J, Zimmermann C, Linzenbold W, Ott G, Enderle M, Albert JG. Bile duct tissue acquisition by cholangioscopy-guided cryobiopsy technique: first-in-human application. VideoGIE. 2023 Feb 15;8(4):158-161. doi: 10.1016/j.vgie.2022.12.007. eCollection 2023 Apr. PMID 37095838
- [Background] Franke KJ, Theegarten D, Hann von Weyhern C, Nilius G, Brueckner C, Hetzel J, Hetzel M, Ruhle KH, Enderle MD, Szyrach MN. Prospective controlled animal study on biopsy sampling with new flexible cryoprobes versus forceps: evaluation of biopsy size, histological quality and bleeding risk. Respiration. 2010;80(2):127-32. doi: 10.1159/000287251. Epub 2010 Feb 17. PMID 20160432
- [Background] Thiboutot J, Illei PB, Maldonado F, Kapp CM, DeMaio A, Lee HJ, Feller-Kopman D, Lentz RJ, Sathyanarayan P, Rahman NM, Silvestri GA, Yarmus L; Interventional Pulmonary Outcomes Group. Safety and Feasibility of a Sheath Cryoprobe for Bronchoscopic Transbronchial Biopsy: The FROSTBITE Trial. Respiration. 2022;101(12):1131-1138. doi: 10.1159/000526876. Epub 2022 Oct 20. PMID 36265451
- [Background] Thompson CC, Kumar N, Slattery J, Clancy TE, Ryan MB, Ryou M, Swanson RS, Banks PA, Conwell DL. A standardized method for endoscopic necrosectomy improves complication and mortality rates. Pancreatology. 2016 Jan-Feb;16(1):66-72. doi: 10.1016/j.pan.2015.12.001. Epub 2015 Dec 22. PMID 26748428
- [Background] Seifert H, Biermer M, Schmitt W, Jurgensen C, Will U, Gerlach R, Kreitmair C, Meining A, Wehrmann T, Rosch T. Transluminal endoscopic necrosectomy after acute pancreatitis: a multicentre study with long-term follow-up (the GEPARD Study). Gut. 2009 Sep;58(9):1260-6. doi: 10.1136/gut.2008.163733. Epub 2009 Mar 11. PMID 19282306
- [Background] Gardner TB, Coelho-Prabhu N, Gordon SR, Gelrud A, Maple JT, Papachristou GI, Freeman ML, Topazian MD, Attam R, Mackenzie TA, Baron TH. Direct endoscopic necrosectomy for the treatment of walled-off pancreatic necrosis: results from a multicenter U.S. series. Gastrointest Endosc. 2011 Apr;73(4):718-26. doi: 10.1016/j.gie.2010.10.053. Epub 2011 Jan 14. PMID 21237454
- [Background] Ramai D, McEntire DM, Tavakolian K, Heaton J, Chandan S, Dhindsa B, Dhaliwal A, Maida M, Anderloni A, Facciorusso A, Adler DG. Safety of endoscopic pancreatic necrosectomy compared with percutaneous and surgical necrosectomy: a nationwide inpatient study. Endosc Int Open. 2023 Apr 4;11(4):E330-E339. doi: 10.1055/a-1994-6214. eCollection 2023 Apr. PMID 37025154
- [Background] Yasuda I, Nakashima M, Iwai T, Isayama H, Itoi T, Hisai H, Inoue H, Kato H, Kanno A, Kubota K, Irisawa A, Igarashi H, Okabe Y, Kitano M, Kawakami H, Hayashi T, Mukai T, Sata N, Kida M, Shimosegawa T. Japanese multicenter experience of endoscopic necrosectomy for infected walled-off pancreatic necrosis: The JENIPaN study. Endoscopy. 2013 Aug;45(8):627-34. doi: 10.1055/s-0033-1344027. Epub 2013 Jun 27. PMID 23807806
- [Background] Yarmus L, Akulian J, Gilbert C, Illei P, Shah P, Merlo C, Orens J, Feller-Kopman D. Cryoprobe transbronchial lung biopsy in patients after lung transplantation: a pilot safety study. Chest. 2013 Mar;143(3):621-626. doi: 10.1378/chest.12-2290. PMID 23328889
- [Background] Pajares V, Puzo C, Castillo D, Lerma E, Montero MA, Ramos-Barbon D, Amor-Carro O, Gil de Bernabe A, Franquet T, Plaza V, Hetzel J, Sanchis J, Torrego A. Diagnostic yield of transbronchial cryobiopsy in interstitial lung disease: a randomized trial. Respirology. 2014 Aug;19(6):900-6. doi: 10.1111/resp.12322. Epub 2014 Jun 1. PMID 24890124